CLINICAL TRIAL: NCT03097315
Title: Open-label Safety Study of Suprachoroidal Triamcinolone Acetonide Injectable Suspension in Patients With Non-Infectious Uveitis
Brief Title: Suprachoroidal Injection of CLS-TA in Patients With Non-infectious Uveitis
Acronym: AZALEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLS1001-302
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Uveitis; Uveitis, Posterior; Uveitis, Anterior; Uveitis, Intermediate; Panuveitis
Keywords: Uveitis; UME; Posterior Uveitis; Anterior Uveitis; Intermediate Uveitis; Panuveitis; Non-infectious Uveitis; Triamcinolone; Choroid; Choroidal Injection; Suprachoroidal; Microneedle; Microinjection; Triamcinolone acetonide
MeSH Terms: conditions — Uveitis; Uveitis, Posterior; Uveitis, Anterior; Uveitis, Intermediate; Panuveitis | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 4 mg CLS-TA Suprachoriodal Injection (Experimental): Suprachoroidal injection of 40 mg/mL (4 mg in 100 μL) of CLS-TA
  Interventions: Drug: 4 mg CLS-TA Suprachoriodal Injection

INTERVENTIONS:
Drug: 4 mg CLS-TA Suprachoriodal Injection — CLS-TA, 40 mg/mL (4 mg in 100 microliters), will be administered as a single injection at 2 timepoints
  Other Names: Triamcinolone Acetonide

SUMMARY:
This open-label study is designed to evaluate the safety of suprachoroidally administered triamcinolone acetone injectable suspension, CLS-TA, in patients with non-infectious uveitis with and without macular edema.

DETAILED DESCRIPTION:
This is a Phase 3, open-label multicenter study to assess the safety of 4 mg of CLS-TA administered via suprachoroidal injection in the treatment of patients diagnosed with noninfectious uveitis with and without macular edema.

Qualified patients will be enrolled and receive two suprachoroidal injections of CLS-TA administered to the study eye approximately 12 weeks apart (Visit 2 and Visit 5). Follow-up visits will be conducted monthly up to 24 weeks (Visit 8).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active or inactive non-infectious uveitis (pan, anterior, intermediate and posterior)
* ETDRS BCVA score of ≥ 5 letters read in the study eye

Exclusion Criteria:

* Any active ocular disease or infection in the study eye other than uveitis
* Intraocular pressure > 22 mmHg or uncontrolled glaucoma in the study eye; patients with IOP of 22 or less in the study eye not excluded with no more than 2 IOP-lowering medications.
* Any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study
* Any topical ocular corticosteroid in the 10 days prior to baseline; intraocular or periocular corticosteroid injections in the 2 months prior to baseline; an OZURDEX implant in the 6 months prior to baseline; RETISERT or ILUVIEN implant in the 3 years prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ciulla, MD, Study Director — Clearside Biomedical, Inc.
Locations (10):
- United States (10):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Northern California Retina Vitreous Associates Medical Group, Inc., Mountain View, California
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Marietta Eye Clinic, Marietta, Georgia
  - Midwest Eye Retina Practicing at Midwest Eye Institute, Indianapolis, Indiana
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jabs DA, Nussenblatt RB, Rosenbaum JT; Standardization of Uveitis Nomenclature (SUN) Working Group. Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop. Am J Ophthalmol. 2005 Sep;140(3):509-16. doi: 10.1016/j.ajo.2005.03.057. PMID 16196117
- [Background] Nussenblatt RB, Palestine AG, Chan CC, Roberge F. Standardization of vitreal inflammatory activity in intermediate and posterior uveitis. Ophthalmology. 1985 Apr;92(4):467-71. doi: 10.1016/s0161-6420(85)34001-0. PMID 4000641
- [Background] Lowder C, Belfort R Jr, Lightman S, Foster CS, Robinson MR, Schiffman RM, Li XY, Cui H, Whitcup SM; Ozurdex HURON Study Group. Dexamethasone intravitreal implant for noninfectious intermediate or posterior uveitis. Arch Ophthalmol. 2011 May;129(5):545-53. doi: 10.1001/archophthalmol.2010.339. Epub 2011 Jan 10. PMID 21220619
- [Derived] Yeh S, Ciulla T. Suprachoroidal triamcinolone acetonide injectable suspension for macular edema associated with noninfectious uveitis: an in-depth look at efficacy and safety. Am J Manag Care. 2023 Feb;29(2 Suppl):S19-S28. doi: 10.37765/ajmc.2023.89324. PMID 36787524
- [Derived] Yeh S, Henry CR, Kapik B, Ciulla TA. Triamcinolone Acetonide Suprachoroidal Injectable Suspension for Uveitic Macular Edema: Integrated Analysis of Two Phase 3 Studies. Ophthalmol Ther. 2023 Feb;12(1):577-591. doi: 10.1007/s40123-022-00603-x. Epub 2022 Nov 18. PMID 36399237

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection
Started | 38
Intention-to-Treat Population (Defined as all patients eligible to be treated with CLS-TA (i.e., patients who did not fail screening and entered the study).) | 38
Safety Population (Defined as all patients who entered the study and were administered at least one dose of CLS-TA.) | 38
Completed | 37
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population included all patients who entered the study and were administered at least one dose of CLS-TA
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants] — Age of patients in years relative to the date of the Screening visit.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 25
    >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of patients in years relative to the date of the Screening visit.
  years | 52.4 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38
Type of Uveitis in the Study Eye [Count of Participants; unit: Participants] — Location of inflammation in the study eye, including anterior (anterior chamber), intermediate (vitreous), posterior (retina or choroid) and panuveitis.
  Participants
    Anterior uveitis | 12
    Intermediate uveitis | 15
    Posterior uveitis | 10
    Panuveitis | 10

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of patients with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs). An adverse event (AE) is the development of an undesirable medical condition or the deterioration of a preexisting medical condition after or during exposure to a pharmaceutical product, whether or not considered causally related to the product. A TEAE is an AE occurring on or after the date of the first dose of study drug or worsening relative to the pre-treatment state. An SAE is an AE that fulfils one or more of the following: results in death; is immediately life-threatening; requires hospitalization nor prolongation of hospitalization; results in persistent or significant disability or incapacity; results in a congenital abnormality or birth defect; or is an important medical event that may jeopardize the subject or may require medical intervention to present one of the outcomes listed above.
Time Frame: Baseline to 24 weeks
Population: The Safety Population included all patients who entered the study and were administered at least one dose of CLS-TA
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection
Number analyzed (Participants) | 38
Participants
  Treatment-Emergent Adverse Events | 27
  Serious Adverse Events | 1

2. Secondary Outcome: Mean Intraocular Pressure in the Study Eye
Description: Intraocular pressure is the fluid pressure inside the eye. Tonometry is the method eye care professionals use to determine this. IOP is an important aspect in the evaluation of patients at risk of glaucoma. Tonometers in this study were calibrated to measure pressure in millimeters of mercury.
Time Frame: Baseline, 24 Weeks
Population: The Safety Population included all patients who entered the study and were administered at least one dose of CLS-TA
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection
Number analyzed (Participants) | 38
mmHg
  Baseline | 13.3 (3.57)
  Week 24 | 15.2 (4.40)

3. Secondary Outcome: Number of Patients With a Grade of 0 in Anterior Chamber Cells in the Study Eye
Description: The anterior chamber is the aqueous humor-filled space inside the eye between the iris and the cornea's innermost surface, the endothelium. The grading of cellular reaction in the anterior chamber helps in the assessment of the severity of uveitis. In this study, anterior chamber cells were graded following the Standardization of Uveitis Nomenclature working group recommendations. The following scale was used to grade the cells in the field: 0 = <1, 0.5+ = 1-5, 1+ = 6-15, 2+ = 16-25, 3+ = 26-50, and 4+ = >50 cells. A lower grade represents less inflammation in the eye.
Time Frame: Baseline, 24 Weeks
Population: The Safety Population included all patients who entered the study and were administered at least one dose of CLS-TA
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection
Number analyzed (Participants) | 38
Participants
  Baseline | 17
  Week 24 | 31

4. Secondary Outcome: Number of Patients With a Grade of 0 in Anterior Chamber Flare in the Study Eye
Description: The anterior chamber is the aqueous humor-filled space inside the eye between the iris and the cornea's innermost surface, the endothelium. The grading of intraocular inflammation or flare in the anterior chamber helps in the assessment of the severity of uveitis. In this study, anterior chamber flare was graded following the Standardization of Uveitis Nomenclature working group recommendations. The following scale was used to grade the flare: 0 = none, 1+ = faint, 2+ moderate (iris and lens details clear), 3+ = marked (iris and lens details hazy), 4+ = intense (fibrin or plastic aqueous). A lower grade represents less inflammation in the eye.
Time Frame: Baseline, 24 Weeks
Population: The Safety Population included all patients who entered the study and were administered at least one dose of CLS-TA
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection
Number analyzed (Participants) | 38
Participants
  Baseline | 27
  Week 24 | 34

5. Secondary Outcome: Number of Patients With a Grade of 0 in Vitreous Haze in the Study Eye
Description: The vitreous body is that part of the eye that fills the space in the center of the eye. The primary purpose of the vitreous body is to keep the center of the eye clear so that light can get to the retina and vision can begin. Vitreous haze involves the obstruction of the back of the eye by vitreous cells and protein exudation. In this study, vitreous haze was graded following a standardized photographic scale ranging from 0 to 4. The following scale was used to grade the vitreous haze: 0 = no inflammation, +0.5 = trace inflammation, +1 = mild blurring of the retinal vessels and optic nerve, +1.5 = optic nerve head and posterior retina view obscuration greater than +1 but less than +2, +2 = moderate blurring of the optic nerve head, +3 = marked blurring of the optic nerve head, +4 = optic nerve head not visible. A lower grade represents less inflammation in the eye.
Time Frame: Baseline, 24 Weeks
Population: The Safety Population included all patients who entered the study and were administered at least one dose of CLS-TA
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection
Number analyzed (Participants) | 38
Participants
  Baseline | 17
  Week 24 | 34

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 24 weeks of follow-up.
Description: Treatment-emergent adverse events were defined as any adverse event occurring on or after the first dose of study drug or worsening from the pre-dose state.
Arm/Group | 4 mg CLS-TA Suprachoriodal Injection
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 1/38
Other Adverse Events (participants affected / at risk) | 24/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 mg CLS-TA Suprachoriodal Injection (N=38)
Visual acuity reduced (Eye disorders) | 1 (1) — # Fellow eye
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 mg CLS-TA Suprachoriodal Injection (N=38)
Conjunctival haemorrhage (Eye disorders) | 5 (5) — # Study eye
Eye inflammation (Eye disorders) | 2 (2) — # Study eye
Eye inflammation (Eye disorders) | 2 (2) — # Fellow eye
Eye pain (Eye disorders) | 3 (5) — # Study eye
Ocular hypertension (Eye disorders) | 2 (3) — # Study eye
Visual acuity reduced (Eye disorders) | 2 (2) — # Study eye
Cataract (Eye disorders) | 2 (2) — # Fellow eye
Cataract nuclear (Eye disorders) | 2 (2) — # Study eye
Cystoid macular oedema (Eye disorders) | 2 (2) — # Fellow eye
Eye irritation (Eye disorders) | 2 (2) — # Fellow eye
Vision blurred (Eye disorders) | 2 (2) — # Fellow eye
Visual impairment (Eye disorders) | 2 (2) — # Fellow eye
Intraocular pressure increased (Investigations) | 4 (4) — # Study eye
Intraocular pressure increased (Investigations) | 4 (4) — # Fellow eye
Procedure headache (Injury, poisoning and procedural complications) | 3 (4) — # Study eye
Injection site pain (General disorders) | 2 (3) — # Study eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institutions and Investigators participating in this study shall have no right to publish or present the results of this study without the prior written consent of Clearside Biomedical, Inc.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT03097315/Prot_SAP_000.pdf